CLINICAL TRIAL: NCT06940583
Title: Comparison of Virtual Reality and Podcast in Improving Patient Experience During Colposcopy: A Randomized Controlled Trial
Brief Title: Comparison of Virtual Reality and Podcast in Improving Patient Experience During Colposcopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinem Ceylan (Other)
Responsible Party: Sponsor-Investigator, Sinem Ceylan, Ankara Medipol University, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VR24
Record Dates: First submitted 2025-04-09; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Stress; Anxiety; Pain; Colposcopy
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): Participants in this group will not receive any distraction during colposcopy. Only standard colposcopy information will be given.
- Podcast (Experimental): Participants will listen to a podcast of relaxing or informative content for 5 minutes before and during colposcopy. Content is based on individual preferences
  Interventions: Other: Podcast
- VR (Experimental): Participants will view a relaxing virtual environment (e.g. nature landscapes, lightly animated themes) for 5 minutes prior to the colposcopy procedure and during the colposcopy wearing a VR headset.
  Interventions: Other: VR

INTERVENTIONS:
Other: VR — Participants will view a relaxing virtual environment (e.g. nature landscapes, lightly animated themes) for 5 minutes prior to the colposcopy procedure and during the colposcopy wearing a VR headset.
  Arms: VR
Other: Podcast — Participants will listen to a podcast of relaxing or informative content for 5 minutes before and 5 minutes during colposcopy. The content will be selected according to individual preferences (e.g. storytelling, humorous content or educational content).
  Arms: Podcast

SUMMARY:
This study wants to see if two things-virtual reality (VR) and podcasts-can help women feel better during a medical test called colposcopy. The study looks at stress, anxiety, pain, and heartbeat. It also checks if women are happy with the test and how long the test takes.

There are three groups: one uses VR, one listens to a podcast, and one gets no extra help.

The study will include 75 women in Turkey. All women are 25 to 65 years old and need to have a colposcopy.

Some women cannot join the study-for example, if they are pregnant, cannot see or hear well, or take strong medicine for pain or stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for colposcopy procedure due to suspicion of cervical squamous intraepithelial lesions.
* Individuals who agree to sign the informed consent form and are willing to participate after being informed about the procedure.
* Individuals who are deemed suitable for the colposcopy procedure and whose health status does not constitute an obstacle to perform this procedure (no visual or hearing impairment).
* Volunteers who speak Turkish at a level to understand the methods and questionnaires used in the study.

Exclusion Criteria:

* Those with claustrophobia, epilepsy, or any other neurological or psychological disorder that may cause discomfort when using the VR headset.
* Individuals with hearing loss that affects their ability to hear podcast content.
* Individuals with vision loss that affects their ability to see VR content.
* Individuals who have previously experienced discomfort while using VR or are unable to adapt to VR
* Individuals who are not suitable for the colposcopy procedure or have a serious health condition that may affect the procedure
* Individuals who are pregnant.
* Individuals with language barriers who may have difficulty understanding the study procedures or distractions.
* Individuals with regular use of sedative or pain medication that may affect stress or pain management during the study.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Before and after colposcopy at 5 min.
  Developed by Cohen, Kamarck and Mermelstein (20) in 1983. PSS was first developed as a 14-item scale and has two other forms, 10 and 4 items. The scale was adapted to Turkish by Eskin et al. PSS was developed to measure the level of stress an individual perceives certain situations as. Participants evaluate the items on a 5-point Likert-type scale.
State Anxiety Inventory | Before and after colposcopy procedure 5 min.
  This scale, developed by Spielberger and his colleagues, consists of two subscales, trait and state, each consisting of 20 questions. The state anxiety scale measures how an individual feels at a certain moment and under certain conditions, while the trait anxiety scale determines how an individual feels regardless of the situation and conditions they are in. The score obtained from the reversed statements is subtracted from the score obtained from the direct statements, and 50 is added to the resulting number for the state anxiety scale and 35 for the trait anxiety scale. The scores obtained from both scales vary between 20-80. As the score obtained from the scale increases, it is evaluated that the person's anxiety level is also high. The adaptation of the scale to Turkish, its validity and reliability study were conducted by Öner and Le Compt
Visual Analog Scale | Before and after colposcopy procedure 5 min.
  The most commonly used and simplest scale. The scale includes numbers between 0-10, where "0" represents no pain and "10" represents the most severe pain. It is an easy-to-understand scale.

SECONDARY OUTCOMES:
Patient Satisfaction Scale | 5 minutes after colposcopy procedure
  "Would you rate your overall satisfaction during the colposcopy procedure on a scale of 0 to 10?" will be asked (0: Not satisfied at all - 10: Very satisfied)
Pulse measurement | 5 minutes before and after the colposcopy procedure.
Prosedur duration | During the colposcopy procedure (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Sinem Ceylan, Study Chair — Ankara Medipol University,Turkey; Özgün Ceylan, Principal Investigator — Etlik City Hospital,Ankara,Turkey; Vakkas Korkmaz, Study Director — Etlik City Hospital,Ankara,Turkey; Gülten Güvenç, Study Chair — Turkey Health Science University,Gulhane Nursing Faculty, Ankara,Turkey; Şahin Kaan Baydemir, Study Chair — Etlik City Hospital,Ankara,Turkey
Locations (1):
- Etlik City Hospital,Department of Gynecology Oncology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No